CLINICAL TRIAL: NCT01483664
Title: Communication Skills Intervention to Promote Transition Into Survivorship
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Maimonides Medical Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Rutgers University (Other); Tampa General Hospital (Other); University of California, Los Angeles (Other); National Cancer Institute (NCI) (NIH); Monash University (Other); Weill Cornell Medical College in Qatar (Other); New York Presbyterian Brooklyn Methodist Hospital (Other); San Francisco State University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-180
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin's Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: patient outcomes; Survivorship; Communication Skills; Communication strategies; Physicians communication; 11-180
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- initial survivorship planning consultation: The overall design follows a cluster-randomized, clinical trial design. Although an apparently statistically-efficient design would have us randomize patients, the CST intervention must be delivered to physicians at four participating sites (MSKCC, Maimonides, MD Anderson, and Moffitt/TGH). Therefore, participating sites will be stratified by size and randomized to either experimental (initial survivorship planning consultation) or control (initial wellness rehabilitation consultation) in a multiple-level, cluster-randomized design, which protects against physician contamination of the experimental intervention within any site.
- initial wellness rehabilitation consultation: The overall design follows a cluster-randomized, clinical trial design. Although an apparently statistically-efficient design would have us randomize patients, the CST intervention must be delivered to physicians at four participating sites (MSKCC, Maimonides, MD Anderson, and Moffitt/TGH). Therefore, participating sites will be stratified by size and randomized to either experimental (initial survivorship planning consultation) or control (initial wellness rehabilitation consultation) in a multiple-level, cluster-randomized design, which protects against physician contamination of the experimental intervention within any site.

SUMMARY:
The purpose of this study is to improve the communication skills of physicians who transition lymphoma cancer patients from the end of treatment to survivorship.

ELIGIBILITY:
Inclusion Criteria:

Physicians:

* who treat patients with DLBCL and HD as per self report

Patients of Physicians:

* have a new diagnosis of Hodgkin's or Diffuse Large B-cell Lymphoma as per pathology report or physician assessment in medical record and/or clinical judgment of the treating physician treated with curative intent.

For part 1 - have scans indicating remission and completing planned chemotherapy and/or radiation therapy. The treating physician will determine that clinical remission has been achieved based on their best judgment.

For part 2 (longitudinal phase): - have new scans indicating remission and completing planned chemotherapy and/or radiation therapy. The treating physician will determine that clinical remission has been achieved based on their best judgment.

* be at least 18 years old
* speak English well enough, in the judgment of the consenting professional, to be able to understand all aspects of the study, provide informed consent, and be able to complete all study measures.

Exclusion Criteria:

Physicians:

* who do not have adequate patients in their clinical practice to meet the 8 patient enrollment requirement for patients with either DLBCL or HD as per self report

Patients of Physicians:

* show evidence of cognitive impairment severe enough to preclude giving permission to the study staff, or completing the survey instruments of the study.
* as per physician judgment, patient's prognosis and/or co-morbidities make them inappropriate for participation in a survivorship study.

For Part 2 ONLY (longitudinal phase):

* those who consented to part 1, consult recording, of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients:
  Patients from each site will be recruited from their respective lymphoma services.
  Physicians:
  Physicians from each site will be recruited from their respective lymphoma services.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2011-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
impact on patient outcomes of targeted physician communication skills training | 3 years

SECONDARY OUTCOMES:
impact of a targeted CST intervention on the physicians | 3 years
  use of strategies, tasks and skills about transitioning lymphoma patients from the end of primary treatment to survivorship.
describe communication during doctor-patient visits during the patients' first three years of survivorship | 3 years
  (MSKCC and MD Anderson baseline data only) The study team will look for qualitative themes to better understand the content of these conversations and the need for survivorship care planning. Half of these recordings were with MSKCC patients and physicians and half were with MD Anderson patients and physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Parker, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Parker PA, Banerjee SC, Matasar MJ, Bylund CL, Franco K, Li Y, Levin TT, Jacobsen PB, Astrow AB, Leventhal H, Horwitz S, Kissane DW. Protocol for a cluster randomised trial of a communication skills intervention for physicians to facilitate survivorship transition in patients with lymphoma. BMJ Open. 2016 Jun 28;6(6):e011581. doi: 10.1136/bmjopen-2016-011581. PMID 27354079
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2015-02-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01483664/ICF_000.pdf